CLINICAL TRIAL: NCT04388969
Title: IIR REGISTRY for the Collection of Real World Data on the Safety and Efficacy of Ambroxol for Patients With Gaucher Disease or GBA Carriers With Parkinson Disease
Brief Title: World Data on Ambroxol for Patients With GD and GBA Related PD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Ari Zimran, Principal Investigator, Shaare Zedek Medical Center
Other Study IDs: 0097-20-SZMC
Record Dates: First submitted 2020-05-10; First posted 2020-05-15 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Gaucher Disease; Parkinson Disease; GBA Gene Mutation
Keywords: Ambroxol; Gaucher Disease; GBA carriers with Parkinson disease
MeSH Terms: conditions — Gaucher Disease; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gaucher disease patients: Patients with type 1,2,3 Gaucher disease.
- GBA carriers with Parkinson disease: Patients with Parkinson disease GBA related (carriers)

SUMMARY:
Ambroxol hydrochloride is an oral mucolytic drug available over-the-counter for many years as cough medicine. In 2009 it was found to also act as a pharmacological chaperone (PC) for mutant glucocerebrosidase, albeit in a several-fold higher dose. Unfortunately, due to its low cost, there have been no pharma-driven clinical trials to establish the use of ambroxol. Thus, data are needed on the safety and efficacy of ambroxol for patients with Gaucher disease (GD).

DETAILED DESCRIPTION:
The three decades of success of enzyme replacement therapy (ERT) for patients with type 1 Gaucher disease (GD1) have been just a partial success to those patients with the more severe neuronopathic forms, particularly the children with myoclonic epilepsy or the infants with type 2 GD.

Ambroxol hydrochloride is an oral mucolytic drug, available over-the-counter (OTC) for many years as cough medicine. In 2009 it was found (in-vitro) to also act as a pharmacological chaperone (PC) for mutant glucocerebrosidase (GCase), albeit in a several-fold higher dose . Unfortunately, due to its low cost, there have been no pharma-driven clinical trials to establish the use of ambroxol.

In an attempt to provide the proof of concept to the potential use of Ambroxol as PC for patients with GD, the Gaucher Clinic at Shaare Zedek Medical Center in Jerusalem, Israel, has treated 12 adult patients with GD1, all untreated with any specific treatment for GD [whether ERT or substrate reduction therapy (SRT),] with Ambroxol at the OTC dose of 150mg/day for a period of 6 months; this was not a formal clinical trial, but rather an audit of a series of patients receiving this drug via the employment of the Israeli Ministry of Health Form 29c to prescribe it for an off-label indication. A single patient, the thinnest of the group with a BMI of 17.1, achieved a robust response relative to baseline similar to ERT.

In 2016, a group from Japan has demonstrated impressive neurological response using high-dose Ambroxol (a marked decrease in seizure frequency, improvement of myoclonus, ability to walk for a bedridden patient, improvement in the latency of I-V waves and threshold of ABR) with dramatic change in daily activities and quality of life (QOL). These encouraging results, that were confirmed in a larger series, yet unpublished, have further led to the conduction of an investigator-initiated-research (IIR) clinical trial in London by Prof A Schapira, which has recently been published (January 13, 2020 JAMA Neurology), wherein newly diagnosed Parkinson patients received high dose Ambroxol, with good safety results

ELIGIBILITY:
Inclusion Criteria:

* patients with Gaucher disease type 1,2 or 3(a,b,c).
* patients with GBA-related Parkinson disease.

Exclusion Criteria:

* None.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Gaucher disease type 1,2,3 (a,b,c) and patients with GBA-related Parkinson disease.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-05-06 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Establishing a registry to be used as a reference for patients,parents and physicians, who consider using Ambroxol | 10 years
  With no specific treatment to offer for patients (particularly children and young adults) with nGD, and with all the above-mentioned encouraging preliminary reports, in our current era of rapidly spreading information (in many meetings worldwide, in the internet and via the social media) individual patients in many countries have started to receive off-label Ambroxol by their treating physicians and a few case reports have been published from Korea , Israel and Canada .
  In order to upscale the level of evidence from anecdotal reports to an observational study, we herein suggest to establish a specific IIR, wherein the "R" stands for a "Registry", that may be used as a reference for patients , parents and physicians, who consider using Ambroxol.
Safety Outcome | 10 years
  By reporting adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ari Zimran, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (2):
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem, Please Select...
  - Shaare Zedek Medical Center, Jerusalem